CLINICAL TRIAL: NCT01433523
Title: Efficacy of ALK House Dust Mite Allergy Immunotherapy Tablet in Subjects With House Dust Mite Induced Asthma. The MITRA Trial
Brief Title: House Dust Mite Treatment of Asthma. The MITRA Trial House Dust Mite Treatment of Asthma
Acronym: MITRA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ALK-Abelló A/S (Industry)
Collaborators: Ergomed (Industry); ACM Pivotal Global Central Laboratory (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MT-04; 2010-018621-19 (EudraCT Number)
Record Dates: First submitted 2011-08-26; First posted 2011-09-14 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Asthma
Keywords: HDM; AIT; asthma; asthma exacerbation; House dust mite induced asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: ALK HDM AIT Placebo
- ALK HDM AIT 6 DU (Experimental)
  Interventions: Drug: ALK HDM AIT 6 DU
- ALK HDM AIT 12 DU (Experimental)
  Interventions: Drug: ALK HDM AIT 12 DU

INTERVENTIONS:
Drug: ALK HDM AIT Placebo — Oral lyophilisate, Placebo, to be administered sublingually once daily
  Arms: Placebo
Drug: ALK HDM AIT 6 DU — Oral lyophilisate, 6 DU, to be administered sublingually once daily for 14-18 months.
  Arms: ALK HDM AIT 6 DU
Drug: ALK HDM AIT 12 DU — Oral lyophilisate, 12 DU, to be administered sublingually once daily for 14-18 months.
  Arms: ALK HDM AIT 12 DU

SUMMARY:
The purpose of this trial is to investigate if treatment with house dust mite allergen immunotherapy tablet can reduce the risk of asthma exacerbation in subjects with house dust mite induced asthma.

ELIGIBILITY:
Key Inclusion Criteria:

* A clinical relevant history consistent with house dust mite induced asthma of at least 1 year prior to trial entry.
* Use of an appropriate amount of inhaled corticosteroid for the control of asthma symptoms.
* Documented reversible airway obstruction.
* Suitable level of asthma control.
* FEV1 ≥ 70% of predicted value.
* Positive Skin Prick Test response to Der pte and/or Der far.
* Positive specific IgE against Der pte and/or Der far (≥ IgE Class 2; ≥ 0.70 KU/L).

Key Exclusion Criteria:

* A clinical history of persistent allergic asthma or rhinitis caused by an allergen to which the subject is regularly exposed and sensitised (except house dust mites).
* A clinical history of intermittent allergic asthma or rhinitis if the seasonal allergen is causing symptoms in the period from October to March.
* Any clinically relevant chronic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 834 (Actual)
Dates: Start 2011-08; Primary Completion 2013-04 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Time to first moderate or severe asthma exacerbation after ICS reduction | Measured during the last 6 months of the trial

SECONDARY OUTCOMES:
Difference in changes in immunological parameters (IgE, IgG4) | Measured at the end of the trial
Time to first severe asthma exacerbation after ICS reduction | Measured during the last 6 months of the trial
Frequency of asthma exacerbations following ICS reduction | Measured during the last 6 months of the trial
The average overall symptom score. | Measured during the last 6 months of the trial
Symptom free days | Measured during the last 6 months of the trial
Number and percentage of subjects with treatment emergent AEs | At end of trial

CONTACTS AND LOCATIONS:
Overall Officials: Christian Virchow, Prof.Dr.med., Principal Investigator — Dept. fof Pneumology, University Clinic Rostock, Ernst-Heydemann-Str. 6, 18057 Rostock, Germany
Locations (1):
- Universitätsklinikum Rostock, Abteilung für Pneumologie Zentrum für Innere Medizin, Ernst Heydemann Strasse 6, Rostock, Germany

REFERENCES:
- [Derived] Hoof I, Bonnelykke K, Stranzl T, Brand S, Li X, Shamji MH, Meyers DA, Bateman ED, Bleecker E, Andersen PS. Genetic and T2 biomarkers linked to the efficacy of HDM sublingual immunotherapy in asthma. Thorax. 2024 Mar 15;79(4):332-339. doi: 10.1136/thorax-2023-220707. PMID 38160049
- [Derived] Fortescue R, Kew KM, Leung MST. Sublingual immunotherapy for asthma. Cochrane Database Syst Rev. 2020 Sep 14;9(9):CD011293. doi: 10.1002/14651858.CD011293.pub3. PMID 32926419